CLINICAL TRIAL: NCT00205452
Title: Does Quality of Life Improve Following Minimally Invasive Parathyroid Surgery?
Brief Title: Quality of Life (QOL) Following Parathyroid Surgery
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2003-164
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Parathyroidectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The only established treatment for the complete resolution of hyperparathyroidism is the surgical removal of the affected glands. While proven as a means of resolving hyperparathyroidism, there have been no comprehensive preoperative and postoperative assessments to determine quality of life for patients undergoing minimally invasive vs. traditional parathyroid surgery. Quality of life will be assessed in subjects undergoing minimally invasive procedures and traditional procedures using a clinically validated survey. We will gather data one week preoperatively as well as one week and one year postoperatively then compare the survey results from the two study groups to each other. We will also compare the study groups to a control group consisting of patients undergoing thyroid surgery. Our ultimate goal is to clarify if minimally invasive parathyroid surgery techniques contribute to a higher patient quality of life as compared to traditional techniques.

ELIGIBILITY:
Inclusion Criteria:

* parathyroidectomy

Exclusion Criteria:

* subjects under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing parathyroid surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2003-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Chen, MD, Principal Investigator — University of Wisconsin Medical School
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States